CLINICAL TRIAL: NCT05018975
Title: Repurposing Tazemetostat for the Treatment of Acute Respiratory Distress Syndrome (ARDS) or Systemic Cytokine Release Syndrome (SCRS) in COVID-19 Patient
Brief Title: Tazemetostat for the Treatment of Moderate to Severe COVID-19 Infection
Acronym: IST
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA recommendation cited safety issues
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2210094
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Cytokine Release Syndrome
Keywords: Systemic Cytokine Release Syndrome Due to SARS-CoV-2 Disease
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — tazemetostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tazemetostat (Experimental): Subjects will receive tazemetostat 800mg BID for 15 days in addition to standard of care treatment. The duration of the interventional part of the study will last 15 days.
  Interventions: Drug: Tazemetostat
- Control (No Intervention): Subjects receiving standard of care treatment

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat 800mg BID PO dosing for 15 days
  Other Names: Tazemetostat oral tablet
  Arms: Tazemetostat

SUMMARY:
The purpose of this study is to assess the safety and efficacy of repurposing tazemetostat for the treatment of Acute Respiratory Distress Syndrome (ARDS) or Systemic Cytokine Release Syndrome (SCRS) in COVID-19 patients.

DETAILED DESCRIPTION:
The investigators hypothesize that tazemetostat will mitigate the hyperinflammatory effects of COVID-19 infection, prevent respiratory deterioration, and reduce requirements of invasive ventilation. This will be conducted as a Phase II open label study. After being informed about the study and potential risks, all patients giving written informed consent will undergo randomization to receive 800 mg tazemetostat BID for 15 days in addition to standard of care treatment. The duration of the interventional part of the study will last 15 days, additionally the patients will be evaluated at 30 and 90 days for overall clinical status and sequelae. The study will be conducted at a single site (Loma Linda University Medical Center).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18-85
* Diagnosed with q-PCR confirmed infection with SARS-Cov-2 virus and admitted to the hospital.
* Receiving non-invasive respiratory support through a nasal cannula or a face mask.
* Ability to take oral medication and be willing to adhere to the tazemetostat regimen.

Exclusion Criteria:

* Unable to take PO medication.
* Need for intubation or ECMO.
* Pregnancy or lactation
* Known allergic reactions to tazemetostat.
* Active malignancy (not in remission).
* Treatment with another investigational drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to one year from date of randomization
  Evaluate the effect of tazemetostat treatment of the course of COVID-19 disease by measuring number of days in hospital from time of randomization to date of discharge or in-hospital death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Ciprian P Gheorghe, MD, PhD, Principal Investigator — Loma Linda University